CLINICAL TRIAL: NCT05020171
Title: Effects of a Lower Limb Strength Training Program on a Seated Robotic Device in Subacute Acquired Brain Injury Patients: a Pilot Study.
Brief Title: Effects of a Lower Limb Strength Training Program on a Seated Robotic Device in Patients
Acronym: Lambda_MIpil
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: many patients missed
Sponsor: Institution de Lavigny (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-00721; 14-O20 (Other Grant/Funding Number: Commission scientifique du domaine santé HES-SO)
Record Dates: First submitted 2021-08-12; First posted 2021-08-25 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: lower limb; robotic device; strength training; subacute; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): group focus on lower limb strength training with a seated robotic device
  Interventions: Device: Group of strength training
- control group (Active Comparator): physiotherapy group as usual, not focused on strength training
  Interventions: Other: Group of physiotherapy not focus on strength training

INTERVENTIONS:
Device: Group of strength training — 2x a week during 5 weeks, strengthening of weak muscles with the intensity recommended in the literature, i.e. 3-4x15 repetition at an intensity of 50 to 80% of the maximum force combined with serious games to stimulate patient involvement in strength training
  Arms: intervention group
Other: Group of physiotherapy not focus on strength training — 2x a week during 5 weeks, active physical therapy treatment based on movement
  Arms: control group

SUMMARY:
The loss of lower limb strength that occurs after an Acquired Brain Injury (ABI) limits the patient's autonomy in participating in activities of daily living, including gait performance. In the sub-acute phase, it is difficult to implement a strengthening program, as weakness prevents exercise being performed with the recommended parameters. This limit can be exceeded by using specific robotic devices, which allow the effort provided to be adapted according to the patient's capacities. In addition, motivation can be improved by the use of feedback or incentive games. The aim of this pilot study is to obtain data on the effect of lower limb strength training with a seated robotic device in subacute ABI patients for a future larger randomised study. In addition, it aims to evaluate the recruitment rate, applicability, resources for implementation and patient tolerance to the training program.

ELIGIBILITY:
Inclusion Criteria:

* Acquired Brain Injury of vascular, traumatic, infectious or tumoral origin in the subacute phase
* Walking ability ≤ Functional Ambulatory Category level 5 (1-6)
* Paresis of the lower limb: strength <57/100 on the Motricity Index
* Cognitive and memory functions allowing the patient to follow treatment instructions and give informed consent

Exclusion Criteria:

* Significant heart problem
* Venous thrombosis less than 6 months
* Musculoskeletal impairment not compatible with movement
* Degenerative neurological disease
* Oxygen-dependent
* Blood pressure not stabilized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
change from study inclusion to end of intervention at 5 weeks in strength of knee extensor's | Study inclusion to end of intervention at 5 weeks
  measure with a manuel dynamometer, in newton

SECONDARY OUTCOMES:
change from study inclusion to end of intervention at 5 weeks in Motricity index legs | Study inclusion to end of intervention at 5 weeks
  clinical manuel strength test, seating on a chair. From 0 to 33, 33 is normal strength.
change from study inclusion to end of intervention at 5 weeks in timed up and go | Study inclusion to end of intervention at 5 weeks
  Mobility test: standing from a chair, walking 3 meters, turn around, returning and seat. in seconds
change from study inclusion to end of intervention at 5 weeks in 10 meters walk test | Study inclusion to end of intervention at 5 weeks
  measure of mean gait speed on 10 meters, at comfortable and maximum gait speed. In meters/second.
change from study inclusion to end of intervention at 5 weeks in Ashworth Scale (spasticity) | Study inclusion to end of intervention at 5 weeks
  measure of the resistance of a muscle to passive stretch according to REsistance to PASsive movement protocol. From 0 to 4, 4 is high spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichonnaz, PhD, Principal Investigator — Haute Ecole de Santé Vaud
Locations (1):
- Institution de Lavigny, Lavigny, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No